CLINICAL TRIAL: NCT07110142
Title: Impact of Tongue Proactive Strengthening Exercise Program on Speech and Swallowing Outcomes Following Partial/Hemiglossectomy and Reconstruction
Brief Title: Tongue Proactive Strengthening Exercise Program Following Partial/Hemi Glossectomy and Reconstruction
Acronym: T-PROSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE6325
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Oral Cancer; Head and Neck Cancer
Keywords: Speech-Language Pathology; Hemiglossectomy; Tongueometer
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Standard of Care(SOC) (No Intervention): Standard of Care (SOC): Standard post-operative care with additional intervention if dysarthria or dysphagia symptoms are not improving as expected
- Arm 2 - SOC + Interventional Group (Experimental): SOC + Interventional Group: Standard post-operative care with biofeedback-driven prophylactic tongue strengthening exercise program using the Tongueometer and the routine interventions if dysarthria or dysphagia symptoms are not improving appropriately
  Interventions: Other: Tongueometer

INTERVENTIONS:
Other: Tongueometer — The Tongueometer device features an air-filled bulb that is placed against the roof of the mouth by the tongue for resistance training. This setup allows for an initial measurement of the patient's maximum tongue strength and endurance, which helps establish goals that are specific to each patient. The device connects to a mobile application that provides visual biofeedback, ensuring consistent monitoring as the patient completes exercises using the tongue bulb for resistance. Once the patient's goals are set based on their initial measurements, the app offers two exercise modules designed to improve both tongue strength and endurance.
  Arms: Arm 2 - SOC + Interventional Group

SUMMARY:
This study is being done to determine whether adding a proactive tongue strengthening exercise program using a biofeedback device (the Tongueometer) improves speech and swallowing outcomes after surgery for tongue cancer. Patients who undergo partial or hemiglossectomy often experience difficulties with speech and swallowing, which can significantly impact their quality of life. While speech and swallow therapy is typically provided in response to problems, this study investigates whether introducing structured tongue strengthening exercises with biofeedback early-can lead to better long-term outcomes. This research will help establish whether this approach should become part of standard post-operative care.

DETAILED DESCRIPTION:
The oral cavity is the most common subsite of head and neck cancers, with over 50,000 new cases diagnosed in 2023 in the United States alone. Of the various anatomic subsites of the oral cavity, the proportion of cancers arising from the tongue is the highest. Surgical resection is the mainstay of treatment and patient may additionally receive chemotherapy and radiation therapy as part of their care. However, removal of a significant portion of the muscular tongue responsible for the complex movements required for speech and swallowing function to obtain negative oncological margins may severely impact function. In recent years, microvascular free flap reconstruction at the time of ablation has become the gold standard to address the oncologic defect and help restore bulk and function to the tongue. In contrast to primary closure or healing by secondary intention, patients who have undergone a resection of a significant portion of their tongue had improved swallowing outcomes in the long term. Despite important restoration of function, however, quality of life and function related to swallowing and speech following reconstruction remain an important problem for some patients. To highlight how important swallowing function is to quality of life, a recent study of hospitalized patients identified tube feed dependence as the sixth debility as equal or worse than death. In addition, severe postoperative dysphagia has been shown to be an independent predictor of overall survival in head and neck cancer patients. This is in addition to post-surgical patients experiencing increased rates of malnutrition, higher number of aspiration events, and decreased speech intelligibility.

Nevertheless, some studies have shown that great functional outcomes can be achieved in the long-term post surgery. Recently, there has been increased effort to identify interventions that are able to improve function in the short and long terms in post-surgical patients. Surgical patients in particular present a challenging patient population, as intervention that is inappropriately early may theoretically increase the risk of peri-operative complications such as wound dehiscence, while delaying therapy may hinder the patient's ability to recover optimal post-operative function. A recent meta-analysis by Lam et al. described a total of eight studies suggesting that as a whole, early interventions increase speech, swallowing function and quality of life in the short term. However, by their own accord the type, duration and start point of the interventions vary greatly among the various studies, and there was significant heterogeneity among the oral subsites of the primary tumor that were included in each study.

Among the studies described, four limit their analyses to tongue resections. The largest of the four studies identified 134 tongue cancer patient undergoing not only resection, but also reconstruction, and early intervention starting on post-operative day 10 was associated with improved EAT-10 and FACT-HN scores in patients undergoing 10 days of tongue and lip exercises, suggesting improved perceived swallowing ability and quality of life in those having undergone this therapy . In terms of more objective measures of outcomes, a similar study of 100 tongue cancer patients by Hsiang et al demonstrated that early swallow therapy decreased the rates of aspiration events and pneumonia at one and four months post-surgery.

From a speech perspective, a systemic review of speech outcomes in patients who underwent hemiglossectomy with free flap reconstruction identified four studies including a total of 238 patients who were reconstructed using a variety of flaps, including radial forearm (RFFF), latissimus dorsi (LD), rectus abdominis (RAM) or anterolateral thigh (ALT). In the largest of those 4 studies, speech was reported as good in 29.4% of patients (clearly understandable) and acceptable in 52.9% of listeners (understandable only when context is known, requiring frequent repetition), which leaves many patients (17.7%) with unintelligible speech. The speech-specific impact on quality of life was not captured in the studies and there remains a paucity of studies investigating the use of early intervention to improve speech in patients following oncologic tongue surgery.

Despite promising data on the efficacy of speech and swallowing interventions following oncologic and reconstructive surgery of the tongue, long term prospective data remains lacking. More information is needed regarding best practices for type and timing of these interventions. Patients at our institutions are commonly referred to the SLP before and immediately after treatment in order to improve speech and prevent dysphagia. However, this is not necessarily the norm, and patients may often be referred only in response to reported speech and/or swallowing difficulties following treatment in the absence of a unified best-practice protocol for the management of post-surgical speech/swallow function. To address this gap, our study aims to compare the effectiveness of active post-surgical tongue strengthening exercise in improving speech and swallow function in patient with tongue cancer. Effectiveness will be measured using a variety of objective and subjective tools commonly used to report speech and swallow outcomes in the head and neck cancer population.

Head and neck cancer patients at our institution are commonly referred to the Speech Language Pathologist (SLP) before, during, and after cancer treatment to improve speech and swallowing. However, this is not standard at many institutions, and patients may often be referred only in response to symptoms of dysfunction following treatment. This is due to the absence of a high quality, evidence-based best-practice protocol for the management of post-treatment speech and swallow function. To address this gap, our study aims to compare the effectiveness of a proactive post-surgical tongue strengthening exercise program using device biofeedback in improving speech and swallow function in patients with tongue cancer. Effectiveness will be measured using a variety of objective and subjective tools commonly used to report speech and swallowing outcomes in the head and neck cancer population. This work will be critical in demonstrating the value of an evidence-based, device-based home tongue rehabilitation program in improving speech and swallow function for oral cancer patients undergoing cancer surgery and reconstruction. This trial will also provide key data to aid in design of a national multi-institutional clinical trial for this concept, which will have the potential to change the standard of care in how we rehabilitate oral cancer patients locoregionally and nationally.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. No prior history of head and neck cancer
3. No prior history of radiation
4. Planned to undergo resection of ≤50% of the native tongue (partial/hemiglossectomy) with immediate reconstruction, including free flap reconstruction, and with or without neck dissection
5. Sufficiently fluent in written English, French, Spanish or Simplified Chinese to complete the study outcomes questionnaires

Exclusion Criteria:

1. Distant metastasis at enrollment
2. Previously seen and treated by speech and language pathologist for dysphagia or dysarthria for non-head and neck cancer causes
3. Prior head and neck radiation
4. Requires mandibulectomy or >50% resection of native tongue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life patient report outcome (PRO) as assessed by Speech Handicap Index(SHI) | 6 months post-treatment
  The Speech Handicap Index (SHI), a validated, self-administered questionnaire consisting of 30 items that assess the functional and psychosocial impact of speech disorders. Each item is rated on a 5-point Likert scale (0 = never, 1 = almost never, 2 = sometimes, 3 = almost always, 4 = always). Scores from all items are summed to produce a total score ranging from 0 to 120, with higher scores indicating a greater perceived speech handicap.

SECONDARY OUTCOMES:
Quality of life patient report outcome (PRO) as assessed by MD Anderson Dysphagia Inventory (MDADI) | 6 months post-treatment
  MDADI: Using this questionnaire, participants score the severity of their symptoms over the previous 24 hours on a scale of 0 (not present) to 10 (as bad as you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ku, MD, FACS, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic
Locations (1):
- Case Comprehensive Cancer Center, Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No